CLINICAL TRIAL: NCT03072069
Title: Analysis of Autonomic Function During Anesthesia Using Response Surface Model
Status: Completed | Type: Observational
Sponsor: National Central University (Other)
Responsible Party: Principal Investigator, Hsin-Yi Wang, Principal Investigator, National Central University
Other Study IDs: NationalCentralU-RSM
Record Dates: First submitted 2017-02-21; First posted 2017-03-07 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia; Reaction; Autonomic Imbalance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Anesthesia in the modern age is at least a two-drug process consisting of an opioid and a sedative hypnotic (e.g., fentanyl and propofol in combination, among others). Therefore, it is important to understand the interaction pharmacodynamics of these agents as they are used clinically. A good method for visualizing the pharmacodynamic interaction behavior of drug combinations is through response surface models. Unlike traditional isobolograms that represent the concentrations of two agents that combine to produce a single degree of drug effect, response surface models characterize the complete spectrum of interaction between two or more agents for all possible levels of concentration and effect. The investigators try to use the response surface model to evaluate the effect of anesthetic combination of autonomic system.

DETAILED DESCRIPTION:
Spectral analysis of heart rate variability (HRV) is a widely used, noninvasive technique to assess autonomic indexes of neural cardiac control. The presence of low-frequency (LF) and high-frequency (HF) oscillatory rhythms in the variability of the R-R interval (RRI) is well established. To date, it is believed that LF is mediated by the parasympathetic and sympathetic systems, whereas HF is mediated primarily by the parasympathetic system. The current study used HRV in order to characterize autonomic nerve system (ANS) activity in patients before and during stable hypnosis, nociceptive surgical stimulation and (adequate) or light (inadequate) analgesia. These effects may vary with the anesthetic technique used. Despite these previous studies, attempts to derive the relation between anesthetic concentrations and HRV have so far remained inconclusive. Such characterization would provide additional information on the behavior of the ANS during different anesthesic drug level and may lay the basis for the development of new clinical application.

Propofol is now widely used in clinical practice because of its favorable recovery profile and low incidence of side effects. However, induction of anesthesia with propofol is often associated with a significant decrease in arterial blood pressure and heart rate (HR). The hypotensive effect of propofol has been attributed to a decrease in systemic vascular resistance or in cardiac output caused by a combination of venous and arterial vasodilation, impaired baroreflex mechanisms and depression of myocardial contractility. Besides, there are some conflicting data regarding the effects of propofol on cardiac sympathetic or parasympathetic tone.

The investigators hypothesis was that at different propofol anesthetic drug level would have reproducible effects on HRV. In addition, these results should be reliably characterized in anesthetized patients provided that HRV uses analysis that can assess transient and rapid changes in ANS activity. Therefore, the first goal of this study was to test the hypothesis that propofol anesthesia would affect HRV depending on the concentrations, and so do opioid and midazolam. Second, the investigators will evaluate the effect of anesthetic combination of autonomic system.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) physical status I who underwent elective surgery.

Exclusion Criteria:

* recent administration of sedative or opioid drugs, emergency surgery and impairment of renal, hepatic, cardiac or respiratory function. No sedative or opioid drugs were administered before induction of anaesthesia.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A prospective, observational, non-randomized study was conducted in 30 patients with American Society of Anaesthesiologists (ASA) physical status I who underwent elective surgery. Participants ages ranged from 20 to 60 years. Exclusion criteria were recent administration of sedative or opioid drugs, emergency surgery and impairment of renal, hepatic, cardiac or respiratory function. No sedative or opioid drugs were administered before induction of anaesthesia.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
change of heart rate variability | up to 24 weeks
  propofol anesthesia or combination with other anesthetics would affect HRV depending on the concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Kun Ting, PhD, Study Director — National Yang Ming Chiao Tung University
Locations (1):
- Department of Surgery, Hsin-chu Branch, Taipei Veterans General Hospital, Taiwan, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
If individual participant data collected in this study are to be made available to other researchers after the end of the study, vital signs and heart rate variability are to be shared, when data will be available.